CLINICAL TRIAL: NCT01024920
Title: A Randomised, Open Label, Parallel Group Phase II Study Comparing the Efficacy and Tolerability of BIBF 1120 Versus Sunitinib in Previously Untreated Patients With Renal Cell Cancer
Brief Title: Compare Safety and Efficacy of BIBF 1120 Versus Sunitinib.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.26; 2009-009516-44 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2009-12-03 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — nintedanib; Sunitinib

ARMS (2):
- Nintedanib (BIBF 1120) (Experimental): Non-marketed substance: Twice daily oral doses of 200mg BIBF 1120 given continuously.
  Interventions: Drug: BIBF 1120
- sunitinib (Active Comparator): Marketed substance: Once a day oral doses of 50mg sunitinib given in repeated 6 week cycles: 4 weeks active, 2 weeks rest.
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: BIBF 1120 — VEGF inhibitor
  Arms: Nintedanib (BIBF 1120)
Drug: sunitinib — VEGF inhibitor
  Arms: sunitinib

SUMMARY:
Compare safety and efficacy of BIBF 1120 versus sunitinib in patients with advanced RCC and to investigate the effects of BIBF 1120 on the heart rate (HR) corrected QT interval (QTcF).

ELIGIBILITY:
Inclusion criteria:

1. Patients with unresectable or metastatic Renal Cell Cancer, who have received no previous systemic anti-cancer treatment.
2. Histological-confirmed diagnosis of renal cell cancer with clear cell component.
3. Acceptable renal,liver,cardiovascular,bone marrow and other functions to allow sunitinib/BIBF 1120 treatment.

Exclusion criteria:

1. Patients unable to tolerate Sunitinib/BIBF 1120 treatment
2. Treatment with other investigational drugs or participation in another clinical study within the past 4 weeks before start of therapy or concomitantly with this study.
3. Patients unable to comply with the 1199.26 protocol.
4. Pregnancy or breast feeding.
5. Active alcohol or drug abuse.
6. Women of child bearing potential, or men who are able to father a child, unwilling to use a medically acceptable form of contraception during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-12-16; Primary Completion 2011-11-08 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- University of Pecs Medical School, Dept. of Oncotherapy, Pécs, Hungary
- Poland (2):
  - Ziemia Lubelska Oncological Center, Lublin, Lublin
  - Onco.Cent. - Instit. of Maria Sklodowskiej-Curie, Warsaw
- Romania (3):
  - Military Central Clinical Emergency Hospital, Bucharest
  - Sf. Nectarie Oncology Center, Craiova, Craiova
  - ONCOLAB SRL, Craiova, Craiova
- Ukraine (5):
  - Municipal Establishment Cherkasy Oncology Centre, Cherkasy
  - Bukovynsk State Medical University, Chernivtsi
  - Munic.Instit."City Clin.Hosp.#4" of Dnipro City Council, Dnipropetrovks
  - CI of LRC Lviv Onco.Reg.Treat.&Diag.Cent., Lviv
  - Uzhgorod National University, Oncology Centre, Uzhhorod
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Surrey Cancer Research Institute, Guildford
  - St James's University Hospital, Leeds

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Eisen T, Shparyk Y, Macleod N, Jones R, Wallenstein G, Temple G, Khder Y, Dallinger C, Studeny M, Loembe AB, Bondarenko I. Effect of small angiokinase inhibitor nintedanib (BIBF 1120) on QT interval in patients with previously untreated, advanced renal cell cancer in an open-label, phase II study. Invest New Drugs. 2013 Oct;31(5):1283-93. doi: 10.1007/s10637-013-9962-7. Epub 2013 Apr 27. PMID 23625328
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, 2:1 randomised, parallel-arm comparison of nintedanib versus sunitinib in patients with advanced renal cell cancer (RCC) who had not received prior systemic therapy.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Nintedanib (BIBF 1120): Participants received orally (swallowed) soft gelatine capsules of nintedanib (BIBF 1120) twice daily (bid) starting with a dose of 200 milligram (mg) bid given continuously in 4-week cycles. Nintedanib was to be swallowed unchewed with about 200 milliliter (mL) of water after food intake with a dosing interval of approximately 12 hours. In case of Adverse Events, the dose was to be reduced to 150 mg bid and 100 mg bid, respectively. The dose was continued daily until withdrawal criteria were fulfilled.
- Sunitinib: Participants received orally (swallowed) hard capsule of sunitinib starting with a dose of 50 milligram (mg) once daily (qd). In case of Adverse Events the dose was to be reduced to 37.5 mg once daily and 25 mg once daily, respectively. The daily dosing was performed in 6-week cycles (4 weeks on and 2 weeks off) until withdrawal criteria were fulfilled.
Period: Overall Study
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Started | 67 | 32
Treated | 64 | 32
Completed | 0 | 0
Not Completed | 67 | 32
Not completed — Progressive disease | 47 | 25
Not completed — Adverse Event | 8 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Patient refusal to continue | 4 | 0
Not completed — Other than listed | 5 | 1
Not completed — Not treated | 3 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib | Total
Number analyzed (Participants) | 64 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (9.7) | 55.5 (11.4) | 58.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 44 | 22 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 32 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
QTcF interval baseline values [Mean (Standard Deviation); unit: millisecconds (ms)] — QTcF interval (QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex (ECG interval consisting of Q, R and S wave) to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula) baseline values were measured at -5 minutes (min), at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h of Day -1 (prior to the first dosing of nintedanib (BIBF 1120)). Population: Full analysis set electrocardiogram (FAS-ECG): All patients in the treated set who were treated with nintedanib (BIBF 1120) and had at least 1 time-matched pair of QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex (Q, R and S wave) to the end of the T wave) measurements available from baseline and from either Day 1 or Day 15 of Treatment Cycle 1 (first 4-week cycle). Only participants with non-missing outcomes were included in the analysis.
  millisecconds (ms)
    -5 minutes: number analyzed (Participants) | 63 | 0 | 63
    -5 minutes | 405.2 (19.6) |  | 405.2 (19.6)
    1 hour (h): number analyzed (Participants) | 63 | 0 | 63
    1 hour (h) | 406.0 (20.3) |  | 406.0 (20.3)
    2 h: number analyzed (Participants) | 63 | 0 | 63
    2 h | 405.3 (19.4) |  | 405.3 (19.4)
    3 h: number analyzed (Participants) | 63 | 0 | 63
    3 h | 406.7 (19.4) |  | 406.7 (19.4)
    4 h: number analyzed (Participants) | 61 | 0 | 61
    4 h | 407.0 (17.8) |  | 407.0 (17.8)
    5 h: number analyzed (Participants) | 61 | 0 | 61
    5 h | 407.2 (18.0) |  | 407.2 (18.0)
    6 h: number analyzed (Participants) | 62 | 0 | 62
    6 h | 405.9 (18.3) |  | 405.9 (18.3)
    7 h: number analyzed (Participants) | 61 | 0 | 61
    7 h | 405.4 (19.2) |  | 405.4 (19.2)
    10 h: number analyzed (Participants) | 60 | 0 | 60
    10 h | 406.6 (19.2) |  | 406.6 (19.2)
    12 h: number analyzed (Participants) | 61 | 0 | 61
    12 h | 406.0 (19.2) |  | 406.0 (19.2)

OUTCOME MEASURES:

1. Primary Outcome: Probability Rates of Progression-free Survival at 9 Months
Description: Progression free survival rate at 9 months is the estimated probability of being alive and not having progressive disease at 9 months after randomisation.
  Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria version 1.1 (RECIST v1.1), at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started together with an absolute increase in the sum of the longest diameters of at least 5 mm, or the appearance of one or more new lesions.
  Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication.
Time Frame: At 9 months after randomisation.
Population: Treated set (TS): All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Probability | 0.431 [0.306 to 0.550] | 0.452 [0.274 to 0.614]
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; Test type: Other; p = 0.8531, Normal approximation test — P-value for comparison of Kaplan-Meier estimates at 9 months using normal approximation test (two-sided)

2. Primary Outcome: Time-matched Change From Baseline to Day 15 in QTcF (QT Interval Corrected by the Fridericia Formula) at 0 Hour (h), at 1 h, at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate by the Fridericia formula. Baseline QTcF measurement at time t was defined as the QTcF measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 15 in QTcF at time t was defined as the QTcF measurement following administration of nintedanib on Day 15 obtained at time t minus baseline QTcF measurement at time t. 0 h is 5 min prior to dosing on Day 15.
  Time-matched change from baseline to Day 15 in QTcF was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 0 h,1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib on Day 15 of are reported.
Time Frame: At 5 minutes (min) before the first dose and at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 15. Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Population: Full analysis set electrocardiogram (FAS-ECG): All patients in the treated set who were treated with nintedanib (BIBF 1120) and had at least 1 time-matched pair of QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex (Q, R and S wave) to the end of the T wave) measurements available from baseline and from either Day 1 or Day 15 of Treatment Cycle 1 (first 4-week cycle). Only participants with non-missing outcomes were included in the analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched change from baseline to Day 15 at -5 minutes (min): number analyzed (Participants) | 63
  Time-matched change from baseline to Day 15 at -5 minutes (min) | 2.6 [-0.7 to 5.9]
  Time-matched change from baseline to Day 15 at 1 hour (h): number analyzed (Participants) | 62
  Time-matched change from baseline to Day 15 at 1 hour (h) | 0.4 [-2.8 to 3.7]
  Time-matched change from baseline to Day 15 at 2 h: number analyzed (Participants) | 63
  Time-matched change from baseline to Day 15 at 2 h | -1.7 [-4.9 to 1.6]
  Time-matched change from baseline to Day 15 at 3 h: number analyzed (Participants) | 63
  Time-matched change from baseline to Day 15 at 3 h | -0.5 [-3.8 to 2.8]
  Time-matched change from baseline to Day 15 at 4 h: number analyzed (Participants) | 61
  Time-matched change from baseline to Day 15 at 4 h | -0.5 [-3.8 to 2.8]
  Time-matched change from baseline to Day 15 at 5 h: number analyzed (Participants) | 61
  Time-matched change from baseline to Day 15 at 5 h | 0.3 [-3.0 to 3.6]
  Time-matched change from baseline to Day 15 at 6 h: number analyzed (Participants) | 62
  Time-matched change from baseline to Day 15 at 6 h | 2.2 [-1.1 to 5.5]
  Time-matched change from baseline to Day 15 at 7 h: number analyzed (Participants) | 61
  Time-matched change from baseline to Day 15 at 7 h | 3.1 [-0.2 to 6.4]
  Time-matched change from baseline to Day 15 at 10 h: number analyzed (Participants) | 60
  Time-matched change from baseline to Day 15 at 10 h | 0.1 [-3.2 to 3.4]
  Time-matched change from baseline to Day 15 at 12 h: number analyzed (Participants) | 60
  Time-matched change from baseline to Day 15 at 12 h | 1.6 [-1.7 to 4.9]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) from randomisation to the occurrence of disease progression (by RECIST Version 1.1) or death, whichever occurred first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started together with an absolute increase in the sum of the longest diameters of at least 5 mm, or the appearance of one or more new lesions.
  Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication.
  The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From the start of study until the cut-off date for 3 year efficacy analysis, up to 3 years.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Months | 8.44 [5.59 to 11.10] | 8.38 [5.59 to 13.86]
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; A stratified log-rank test (two-sided, 0.05 significance level) was used to test the effect of nintedanib on PFS compared with sunitinib. The test was stratified by Motzer risk score category (low/intermediate or high) and prior nephrectomy surgery for Renal Cell Cancer (yes or no); Test type: Other; p = 0.6395, Log Rank; Hazard Ratio (HR) = 1.120, 95% CI 2-sided [0.697 to 1.800] — Hazard ratio from Cox proportional hazards model stratified by Motzer risk score and previous surgery

4. Secondary Outcome: Objective Response According to RECIST Criteria
Description: Objective response was defined as complete response (CR, the disappearance of all target and non-target lesions and no new lesions) or partial response (PR, at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters and no new lesions) as determined by RECIST Version 1.1. Numbers of participants with objective response are reported.
  Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication.
Time Frame: From the start of study until the cut-off date for 3 year efficacy analysis, up to 3 years.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Participants
  Complete Response | 0 | 1
  Partial response | 14 | 11
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; A logistic regression model stratified by Motzer risk score category and prior surgery for renal cell cancer (RCC) was used to compare the objective response rate between the two treatment arms. The corresponding odds ratio and 95% Confidence Intervals was also presented; Test type: Other; p = 0.1213, Regression, Logistic; Odds Ratio (OR) = 0.484, 95% CI 2-sided [0.193 to 1.212] — Odds ratio > 1 favours nintedanib

5. Secondary Outcome: Duration of Objective Response
Description: Duration (months) of objective response was measured from the time of first objective response to the time of disease progression (by RECIST Version 1.1) or death, whichever occurred first.
  Objective response was defined as complete response (CR, the disappearance of all target and non-target lesions and no new lesions) or partial response (PR, at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of the longest diameters and no new lesions) as determined by RECIST Version 1.1.
  Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication. The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From the time of first objective response to the time of disease progression or death (whichever comes first), up to 3 years.
Population: Treated set (TS): All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment and showed objective response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 14 | 12
Months | 19.42 [8.31 to NA] — Upper Interquartile-Range cannot be estimated based on the current limited data in a small sample-sized study. | 11.66 [7.06 to 28.45]

6. Secondary Outcome: Overall Survival
Description: Overall survival was calculated as the time (months) from randomisation to death. Patients for whom there was no evidence of death at the time of analysis were censored on the date that they were last known to have been alive.
  The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From randomisation to death, up to 3 years.
Population: Treated Set (TS) : All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Months | 20.37 [13.86 to 29.01] | 21.22 [11.01 to 31.74]
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; Test type: Other; p = 0.7593, Log Rank — P-value from log-rank stratified by Motzer risk score and previous surgery; Hazard Ratio (HR) = 0.920, 95% CI 2-sided [0.542 to 1.564] — Hazard ratio from Cox proportional hazards model stratified by Motzer risk score and previous surgery. Hazard ratio < 1 favours nintedanib

7. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time period from randomisation to objective tumour progression. Patients with no progression (by RECIST Version 1.1) were censored at the date of the last evaluable imaging.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started together with an absolute increase in the sum of the longest diameters of at least 5 mm, or the appearance of one or more new lesions.
  Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication. The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From randomisation up to objective tumour progression, up to 3 years.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Months | 8.48 [7.56 to 11.20] | 8.54 [5.68 to 13.90]
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; Test type: Other; p = 0.5958, Log Rank; P-value from log-rank stratified by Motzer risk score and previous surgery; Cox Proportional Hazard = 1.143, 95% CI 2-sided [0.697 to 1.873] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from randomisation to objective tumour progression (by RECIST Version 1.1), death, global deterioration of health status requiring treatment discontinuation, or start of new anticancer treatment, whichever came first. Tumour imaging was made by investigators using Computed tomography (CT)/Magnetic Resonance imaging (MRI) every 12 weeks after the first administration of the trial medication.The Kaplan-Meier method was used to calculate the estimates.
Time Frame: From randomisation up to objective tumour progression, up to 3 years.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Month | 8.44 [5.62 to 10.97] | 8.36 [5.55 to 13.86]
Statistical Analysis 1: Comparison: Nintedanib (BIBF 1120) vs Sunitinib; Test type: Other; p = 0.5712, Log Rank; P-value from log-rank stratified by Motzer risk score and previous surgery (two-sided); Hazard Ratio (HR) = 1.142, 95% CI 2-sided [0.720 to 1.812] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Time-matched Change From Baseline to Day 1 in QTcF (QT Interval Corrected by the Fridericia Formula) at 1 Hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate by the Fridericia formula. Baseline QTcF measurement at time t was defined as the QTcF measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 in QTcF at time t was defined as the QTcF measurement following administration of nintedanib on Day 1 obtained at time t minus baseline QTcF measurement at time t.
  Time-matched change from baseline to Day 1 in QTcF was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib on Day 1 are reported.
Time Frame: At 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 of treatment Cycle 1. Baseline (Day -1) values were taken at exactly the same time points as on Day 1.
Population: Full analysis set electrocardiogram (FAS-ECG): All patients in the treated set who were treated with nintedanib (BIBF 1120) and had at least 1 time-matched pair of QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) measurements available from baseline and from either Day 1 or Day 15 of Treatment Cycle 1 (first 4-week cycle). Only participants with non-missing outcomes were included in the analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched change from baseline to Day 1 at 1 hour (h) | -1.6 [-4.4 to 1.2]
  Time-matched change from baseline to Day 1 at 2 h | -3.1 [-6.0 to -0.3]
  Time-matched change from baseline to Day 1 at 3 h | -2.6 [-5.5 to 0.2]
  Time-matched change from baseline to Day 1 at 4 h: number analyzed (Participants) | 62
  Time-matched change from baseline to Day 1 at 4 h | -2.6 [-5.4 to 0.3]
  Time-matched change from baseline to Day 1 at 5 h: number analyzed (Participants) | 62
  Time-matched change from baseline to Day 1 at 5 h | -1.4 [-4.3 to 1.4]
  Time-matched change from baseline to Day 1 at 6 h: number analyzed (Participants) | 62
  Time-matched change from baseline to Day 1 at 6 h | -2.0 [-4.8 to 0.9]
  Time-matched change from baseline to Day 1 at 7 h: number analyzed (Participants) | 61
  Time-matched change from baseline to Day 1 at 7 h | -1.5 [-4.4 to 1.3]
  Time-matched change from baseline to Day 1 at 10 h: number analyzed (Participants) | 60
  Time-matched change from baseline to Day 1 at 10 h | -3.6 [-6.4 to -0.7]
  Time-matched change from baseline to Day 1 at 12 h: number analyzed (Participants) | 61
  Time-matched change from baseline to Day 1 at 12 h | -2.2 [-5.0 to 0.7]

10. Secondary Outcome: Time-matched Change From Baseline in QTcF Interval (QT Interval Corrected by the Fridericia Formula) at the Time of Each Participant's Maximum Plasma Concentration of Nintedanib (BIBF 1120), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula. Baseline QTcF measurement at time t was defined as the QTcF measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QTcF at time t was defined as the QTcF measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QTcF measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QTcF' at the time of the participant's maximum nintedanib plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: At 5 minutes (min) before the first dose on Day 15 and at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15 of the first treatment cycle. Continues in the description.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched change from baseline in QTcF interval at maximum BIBF 1120 concentration on Day 1 | -2.8 [-5.0 to -0.6]
  Time-matched change from baseline in QTcF interval at maximum BIBF 1120 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in QTcF interval at maximum BIBF 1120 concentration on Day 15 | -3.2 [-5.9 to -0.4]

11. Secondary Outcome: Time-Matched Change From Baseline in QTcF Interval at the Time of Each Patient's Maximum Plasma Concentration of BIBF 1202 (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Baseline QTcF measurement at time t was defined as the QTcF measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QTcF at time t was defined as the QTcF measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QTcF measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QTcF' at the time of the participant's maximum BIBF 1202 (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched change from baseline in QTcF interval at maximum BIBF 1202 concentration on Day 1: number analyzed (Participants) | 63
  Time-matched change from baseline in QTcF interval at maximum BIBF 1202 concentration on Day 1 | -2.5 [-4.6 to -0.5]
  Time-matched change from baseline in QTcF interval at maximum BIBF 1202 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in QTcF interval at maximum BIBF 1202 concentration on Day 15 | -1.1 [-3.8 to 1.6]

12. Secondary Outcome: Time-Matched Change From Baseline in QTcF Interval at the Time of Each Patient's Maximum Plasma Concentration of BIBF 1202-glucuronide (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Baseline QTcF measurement at time t was defined as the QTcF measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QTcF at time t was defined as the QTcF measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QTcF measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QTcF' at the time of the participant's maximum BIBF 1202-glucuronide (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched change in QTcF from baseline at maximum BIBF 1202-glucuronide concentration on Day 1: number analyzed (Participants) | 60
  Time-matched change in QTcF from baseline at maximum BIBF 1202-glucuronide concentration on Day 1 | -2.4 [-4.9 to 0.0]
  Time-matched change in QTcF from baseline at maximum BIBF 1202-glucuronide concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change in QTcF from baseline at maximum BIBF 1202-glucuronide concentration on Day 15 | -1.5 [-4.2 to 1.2]

13. Secondary Outcome: Average Time-matched Changes From Baseline in QTcF Interval Over 1 h to 12 h After Dosing on Days 1 and 15 of Treatment Cycle 1
Description: Average time-matched in QTcF interval (QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula) changes over 1 to 12 hours was evaluated using a t-test for paired observation. The mean differences between post-treatment values (Days 1 and 15) and baseline (Day -1) along with two-sided 90% confidence limits are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 1 and on Day 15.
Time Frame: At 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15 of first treatment cycle. Continues in the description.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Averaged time-matched changes from baseline in QTcF interval over 1 h to 12 h after dosing on Day 1 | -2.2 [-3.5 to -0.8]
  Averaged time-matched changes from baseline in QTcF interval over 1 h to 12 h after dosing on Day 15: number analyzed (Participants) | 63
  Averaged time-matched changes from baseline in QTcF interval over 1 h to 12 h after dosing on Day 15 | 0.5 [-1.4 to 2.3]

14. Secondary Outcome: Time-matched Changes From Baseline to Day 15 in QT Interval at 0 Hour (h), at 1 h, at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: QT interval is the electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave. Baseline QT measurement at time t was defined as the QT measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 15 in QT at time t was defined as the QT measurement following administration of nintedanib on Day 15 obtained at time t minus baseline QT measurement at time t. 0 h is 5 min prior to dosing on Day 15.
  Time-matched change from baseline to Day 15 in QT was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 0 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib on Day 15 of Cycle 1are reported.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Time-matched QT interval change from baseline to Day 15 at -5 minutes (min): number analyzed (Participants) | 63
  Time-matched QT interval change from baseline to Day 15 at -5 minutes (min) | 1.0 [-3.6 to 5.6]
  Time-matched QT interval change from baseline to Day 15 at 1 hour (h): number analyzed (Participants) | 62
  Time-matched QT interval change from baseline to Day 15 at 1 hour (h) | 0.5 [-4.1 to 5.1]
  Time-matched QT interval change from baseline to Day 15 at 2 h: number analyzed (Participants) | 63
  Time-matched QT interval change from baseline to Day 15 at 2 h | 1.6 [-3.0 to 6.2]
  Time-matched QT interval change from baseline to Day 15 at 3 h: number analyzed (Participants) | 63
  Time-matched QT interval change from baseline to Day 15 at 3 h | 4.4 [-0.2 to 9.0]
  Time-matched QT interval change from baseline to Day 15 at 4 h: number analyzed (Participants) | 61
  Time-matched QT interval change from baseline to Day 15 at 4 h | 4.7 [0.0 to 9.3]
  Time-matched QT interval change from baseline to Day 15 at 5 h: number analyzed (Participants) | 61
  Time-matched QT interval change from baseline to Day 15 at 5 h | 5.1 [0.5 to 9.7]
  Time-matched QT interval change from baseline to Day 15 at 6 h: number analyzed (Participants) | 62
  Time-matched QT interval change from baseline to Day 15 at 6 h | 7.7 [3.1 to 12.3]
  Time-matched QT interval change from baseline to Day 15 at 7 h: number analyzed (Participants) | 61
  Time-matched QT interval change from baseline to Day 15 at 7 h | 7.1 [2.5 to 11.7]
  Time-matched QT interval change from baseline to Day 15 at 10 h: number analyzed (Participants) | 60
  Time-matched QT interval change from baseline to Day 15 at 10 h | 3.4 [-1.2 to 8.0]
  Time-matched QT interval change from baseline to Day 15 at 12 h: number analyzed (Participants) | 60
  Time-matched QT interval change from baseline to Day 15 at 12 h | 4.2 [-0.4 to 8.8]

15. Secondary Outcome: Time-matched Changes From Baseline to Day 1 in QT Interval at 1 Hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: QT interval is the electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave. Baseline QT measurement at time t was defined as the QT measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 in QT at time t was defined as the QT measurement following administration of nintedanib on Day 1 obtained at time t minus baseline QT measurement at time t.
  Time-matched change from baseline to Day 1 in QT was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib on Day 1 are reported.
Time Frame: At 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1. Baseline (Day -1) values were taken at exactly the same time points as on Day 1.
Population: as for outcome 9
Measure: Least Squares Mean (90% Confidence Interval); unit: millisecond (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
millisecond (ms)
  Time-matched QT interval change from baseline to Day 1 at 1 hour (h) | -2.0 [-6.3 to 2.3]
  Time-matched QT interval change from baseline to Day 1 at 2 h | 1.6 [-2.8 to 5.9]
  Time-matched QT interval change from baseline to Day 1 at 3 h | 3.5 [-0.8 to 7.8]
  Time-matched QT interval change from baseline to Day 1 at 4 h: number analyzed (Participants) | 62
  Time-matched QT interval change from baseline to Day 1 at 4 h | 1.4 [-2.9 to 5.7]
  Time-matched QT interval change from baseline to Day 1 at 5 h: number analyzed (Participants) | 62
  Time-matched QT interval change from baseline to Day 1 at 5 h | 1.4 [-2.9 to 5.7]
  Time-matched QT interval change from baseline to Day 1 at 6 h: number analyzed (Participants) | 62
  Time-matched QT interval change from baseline to Day 1 at 6 h | 1.8 [-2.6 to 6.1]
  Time-matched QT interval change from baseline to Day 1 at 7 h: number analyzed (Participants) | 61
  Time-matched QT interval change from baseline to Day 1 at 7 h | 0.7 [-3.6 to 5.0]
  Time-matched QT interval change from baseline to Day 1 at 10 h: number analyzed (Participants) | 60
  Time-matched QT interval change from baseline to Day 1 at 10 h | -1.7 [-6.0 to 2.7]
  Time-matched QT interval change from baseline to Day 1 at 12 h: number analyzed (Participants) | 61
  Time-matched QT interval change from baseline to Day 1 at 12 h | -2.2 [-6.5 to 2.2]

16. Secondary Outcome: Time-Matched Change From Baseline in QT Interval at the Time of Each Patient's Maximum Plasma Concentration of Nintedanib (BIBF 1120), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QT interval is the (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave. Baseline QT measurement at time t was defined as the QT measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QT at time t was defined as the QT measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QT measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QT' at the time of the participant's maximum nintedanib plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 1 and on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: millisecond (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
millisecond (ms)
  Time-matched change from baseline in QT interval at maximum BIBF 1120 concentration on Day 1 | 0.9 [-2.3 to 4.0]
  Time-matched change from baseline in QT interval at maximum BIBF 1120 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in QT interval at maximum BIBF 1120 concentration on Day 15 | -0.4 [-5.0 to 4.1]

17. Secondary Outcome: Time-Matched Change From Baseline in QT Interval at the Time of Each Patient's Maximum Plasma Concentration of BIBF 1202 (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QT interval is the (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave. Baseline QT measurement at time t was defined as the QT measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QT at time t was defined as the QT measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QT measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QT' at the time of the participant's maximum BIBF 1202 (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: At 5 minutes (min) before the first dose on Day 15 and at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15 of first treatment cycle. Continues in the description.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: millisecond (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
millisecond (ms)
  Time-matched change from baseline in QT interval at maximum BIBF 1202 concentration on Day 1: number analyzed (Participants) | 63
  Time-matched change from baseline in QT interval at maximum BIBF 1202 concentration on Day 1 | 1.2 [-1.9 to 4.3]
  Time-matched change from baseline in QT interval at maximum BIBF 1202 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in QT interval at maximum BIBF 1202 concentration on Day 15 | 1.8 [-2.7 to 6.3]

18. Secondary Outcome: Time-Matched Change From Baseline in QT Interval at the Time of Each Patient's Maximum Plasma Concentration BIBF 1202-glucuronide (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QT interval is the (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave. Baseline QT measurement at time t was defined as the QT measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in QT at time t was defined as the QT measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline QT measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in QT' at the time of the participant's maximum BIBF 1202-glucuronide (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: millisecond (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
millisecond (ms)
  Time-matched change from baseline in QT at maximum BIBF 1202-glucuronide concentration on Day 1: number analyzed (Participants) | 60
  Time-matched change from baseline in QT at maximum BIBF 1202-glucuronide concentration on Day 1 | -0.4 [-4.0 to 3.1]
  Time-matched change from baseline in QT at maximum BIBF 1202-glucuronide concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in QT at maximum BIBF 1202-glucuronide concentration on Day 15 | 1.3 [-3.2 to 5.9]

19. Secondary Outcome: Averaged Time-matched Changes From Baseline in QT Interval (Electrocardiogram (ECG) Interval From the Beginning of the QRS Complex to the End of the T Wave) Over 1 h to 12 h After Dosing on Days 1 and 15 of Treatment Cycle 1
Description: Averaged time-matched QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) changes from baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120) to Day 1 (first drug dose nintedanib (BIBF 1120)) and to Day 15 (steady state) over 1 to 12 hours was evaluated using a t-test for paired observation. The mean differences between post-treatment values (Days 1 and 15) and baseline (Day -1) along with two-sided 90% confidence limits are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 1 and on Day 15.
Time Frame: At 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15 of first treatment cycle.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: millisecond (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
millisecond (ms)
  Averaged time-matched changes from baseline in QT interval over 1 h to 12 h after dosing on Day 1 | 0.9 [-1.3 to 3.0]
  Averaged time-matched changes from baseline in QT interval over 1 h to 12 h after dosing on Day 15: number analyzed (Participants) | 63
  Averaged time-matched changes from baseline in QT interval over 1 h to 12 h after dosing on Day 15 | 4.2 [0.6 to 7.7]

20. Secondary Outcome: Time-Matched Heart Rate (HR) Changes From Baseline to Day 15 at 0 Hour (h), at 1 h, at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: Baseline heart rate (HR) measurement at time t was defined as the HR measurement collected 1 day prior to the day of the first administration of nintedanib (BIBF 1120) at time t. Time-matched change from baseline to Day 15 in HR at time t was defined as the HR measurement following administration of nintedanib (BIBF 1120) on Day 15 obtained at time t minus baseline HR measurement at time t. 0 h is 5 min prior to dosing on Day 15.
  Time-matched change from baseline to Day 15 in HR was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 0 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib (BIBF 1120) on Day 15 of Cycle 1 are reported.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Time-matched heart rate (HR) change from baseline to Day 15 at -5 minutes (min): number analyzed (Participants) | 63
  Time-matched heart rate (HR) change from baseline to Day 15 at -5 minutes (min) | 0.9 [-1.2 to 3.0]
  Time-matched heart rate (HR) change from baseline to Day 15 at 1 h: number analyzed (Participants) | 62
  Time-matched heart rate (HR) change from baseline to Day 15 at 1 h | -0.3 [-2.4 to 1.9]
  Time-matched heart rate (HR) change from baseline to Day 15 at 2 h: number analyzed (Participants) | 63
  Time-matched heart rate (HR) change from baseline to Day 15 at 2 h | -2.0 [-4.2 to 0.1]
  Time-matched heart rate (HR) change from baseline to Day 15 at 3 h: number analyzed (Participants) | 63
  Time-matched heart rate (HR) change from baseline to Day 15 at 3 h | -3.3 [-5.4 to -1.2]
  Time-matched heart rate (HR) change from baseline to Day 15 at 4 h: number analyzed (Participants) | 61
  Time-matched heart rate (HR) change from baseline to Day 15 at 4 h | -3.4 [-5.5 to -1.3]
  Time-matched heart rate (HR) change from baseline to Day 15 at 5 h: number analyzed (Participants) | 61
  Time-matched heart rate (HR) change from baseline to Day 15 at 5 h | -3.1 [-5.2 to -1.0]
  Time-matched heart rate (HR) change from baseline to Day 15 at 6 h: number analyzed (Participants) | 62
  Time-matched heart rate (HR) change from baseline to Day 15 at 6 h | -3.8 [-5.9 to -1.7]
  Time-matched heart rate (HR) change from baseline to Day 15 at 7 h: number analyzed (Participants) | 61
  Time-matched heart rate (HR) change from baseline to Day 15 at 7 h | -2.8 [-4.9 to -0.7]
  Time-matched heart rate (HR) change from baseline to Day 15 at 10 h: number analyzed (Participants) | 60
  Time-matched heart rate (HR) change from baseline to Day 15 at 10 h | -2.4 [-4.5 to -0.5]
  Time-matched heart rate (HR) change from baseline to Day 15 at 12 h: number analyzed (Participants) | 60
  Time-matched heart rate (HR) change from baseline to Day 15 at 12 h | -1.6 [-3.8 to 0.5]

21. Secondary Outcome: Time-Matched Heart Rate (HR) Changes From Baseline to Day 1 at 1 Hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h After Dosing of Nintedanib (BIBF 1120)
Description: Baseline heart rate (HR) measurement at time t was defined as the HR measurement collected 1 day prior to the day of the first administration of nintedanib (BIBF 1120) at time t. Time-matched change from baseline to Day 1 in HR at time t was defined as the HR measurement following administration of nintedanib (BIBF 1120) on Day 1 obtained at time t minus baseline HR measurement at time t.
  Time-matched change from baseline to Day 1 in HR was modelled using a linear mixed-effects model for repeated measures which included 'time' as repeated measures and the time-matched baseline value as a covariate. Adjusted means with corresponding 2-sided 90% confidence intervals at 0 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 10 h and 12 h after dosing of nintedanib (BIBF 1120) on Day 1 are reported.
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Time-matched heart rate (HR) change from baseline to Day 1 at 1 hour (h) | -0.0 [-1.9 to 1.8]
  Time-matched heart rate (HR) change from baseline to Day 1 at 2 h | -2.9 [-4.7 to -1.0]
  Time-matched heart rate (HR) change from baseline to Day 1 at 3 h | -3.8 [-5.7 to -2.0]
  Time-matched heart rate (HR) change from baseline to Day 1 at 4 h: number analyzed (Participants) | 62
  Time-matched heart rate (HR) change from baseline to Day 1 at 4 h | -2.5 [-4.3 to -0.6]
  Time-matched heart rate (HR) change from baseline to Day 1 at 5 h: number analyzed (Participants) | 62
  Time-matched heart rate (HR) change from baseline to Day 1 at 5 h | -1.8 [-3.7 to 0.0]
  Time-matched heart rate (HR) change from baseline to Day 1 at 6 h: number analyzed (Participants) | 62
  Time-matched heart rate (HR) change from baseline to Day 1 at 6 h | -2.2 [-4.1 to -0.4]
  Time-matched heart rate (HR) change from baseline to Day 1 at 7 h: number analyzed (Participants) | 61
  Time-matched heart rate (HR) change from baseline to Day 1 at 7 h | -1.4 [-3.3 to 0.4]
  Time-matched heart rate (HR) change from baseline to Day 1 at 10 h: number analyzed (Participants) | 60
  Time-matched heart rate (HR) change from baseline to Day 1 at 10 h | -1.3 [-3.2 to 0.6]
  Time-matched heart rate (HR) change from baseline to Day 1 at 12 h: number analyzed (Participants) | 61
  Time-matched heart rate (HR) change from baseline to Day 1 at 12 h | 0.0 [-1.8 to 1.9]

22. Secondary Outcome: Time-Matched Change From Baseline in Heart Rate (HR) at the Time of Each Patient's Maximum Nintedanib (BIBF 1120) Plasma Concentration, Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Baseline heart rate (HR) measurement at time t was defined as the HR measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in HR at time t was defined as the HR measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline HR measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in HR' at the time of the participant's maximum nintedanib plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Time-matched change from baseline in HR at maximum BIBF 1120 concentration on Day 1 | -2.0 [-3.4 to -0.7]
  Time-matched change from baseline in HR at maximum BIBF 1120 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in HR at maximum BIBF 1120 concentration on Day 15 | -2.1 [-4.3 to 0.1]

23. Secondary Outcome: Time-Matched Change From Baseline in Heart Rate (HR) at the Time of Each Patient's Maximum Plasma Concentration of BIBF 1202 (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Baseline heart rate (HR) measurement at time t was defined as the HR measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in HR at time t was defined as the HR measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline HR measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in HR' at the time of the participant's maximum BIBF 1202 (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Time-matched change from baseline in HR at maximum BIBF 1202 concentration on Day 1: number analyzed (Participants) | 63
  Time-matched change from baseline in HR at maximum BIBF 1202 concentration on Day 1 | -2.3 [-3.8 to -0.8]
  Time-matched change from baseline in HR at maximum BIBF 1202 concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in HR at maximum BIBF 1202 concentration on Day 15 | -2.0 [-4.2 to 0.1]

24. Secondary Outcome: Time-Matched Change From Baseline in Heart Rate (HR) at the Time of Each Patient's Maximum Plasma Concentration of BIBF 1202-glucuronide (a Nintedanib (BIBF 1120) Metabolite), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Baseline heart rate (HR) measurement at time t was defined as the HR measurement collected 1 day prior to the day of the first administration of nintedanib at time t. Time-matched change from baseline to Day 1 (Day 15) in HR at time t was defined as the HR measurement following administration of nintedanib on Day 1 (Day 15) obtained at time t minus baseline HR measurement at time t.
  For each participant 'Time-matched change from baseline to Day 1 (Day 15) in HR' at the time of the participant's maximum BIBF 1202-glucuronide (a nintedanib (BIBF 1120) metabolite) plasma concentration was obtained and the mean across all participants calculated. Corresponding two-sided 90% confidence intervals based on the t-distribution are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 1 and on Day 15.
Time Frame: At 5 minutes (min) before the first dose on Day 15 and at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15 of treatment cycle 1. Continues in the description.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Time-matched change from baseline in HR at maximum BIBF 1202-glucuronide concentration on Day 1: number analyzed (Participants) | 60
  Time-matched change from baseline in HR at maximum BIBF 1202-glucuronide concentration on Day 1 | -1.2 [-2.6 to 0.3]
  Time-matched change from baseline in HR at maximum BIBF 1202-glucuronide concentration on Day 15: number analyzed (Participants) | 62
  Time-matched change from baseline in HR at maximum BIBF 1202-glucuronide concentration on Day 15 | -1.6 [-3.6 to 0.4]

25. Secondary Outcome: Averaged Time-Matched Heart Rate (HR) Change From Baseline Over 1 to 12 Hours, Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Averaged time-matched heart rate changes from baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) to Day 1 (first drug dose nintedanib (BIBF 1120)) and to Day 15 (steady state) over 1 to 12 hours was evaluated using a t-test for paired observation. The mean differences between post-treatment values (Days 1 and 15) and baseline (Day -1) along with two-sided 90% confidence limits are reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 1 and on Day 15.
Time Frame: At 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1 and on Day 15.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
beats per minute (bpm)
  Averaged time-matched HR change from baseline over 1 to 12 hours on Day 1 | -1.9 [-2.8 to -1.1]
  Averaged time-matched HR change from baseline over 1 to 12 hours on Day 15: number analyzed (Participants) | 63
  Averaged time-matched HR change from baseline over 1 to 12 hours on Day 15 | -2.5 [-4.0 to -0.9]

26. Secondary Outcome: Frequency of Patients With Maximum Time-Matched QTcF Interval Change From Baseline Categorized by Magnitude of Change, Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula.
  Number of patients with maximum time-matched change from baseline in the QTcF interval observed at each point in time, i.e., 9 time points on Day 1 and 10 timepoints on Day 15 is reported. 3 categories of individual QTcF increases from baseline to maximum value were defined:
  <= 30 milliseconds (ms)
  > 30 to 60 milliseconds (ms)
  > 60 milliseconds (ms) Changes more than 60 ms in the QTcF interval represent notable changes. Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 1, 1-12 hours (h): <= 30 milliseconds (ms) | 64
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 1, 1-12 hours (h): > 30 to 60 milliseconds (ms) | 0
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 1, 1-12 hours (h): > 60 milliseconds (ms) | 0
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: number analyzed (Participants) | 63
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: <= 30 milliseconds (ms) | 57
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: > 30 to 60 milliseconds (ms) | 6
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: > 60 milliseconds (ms) | 0

27. Secondary Outcome: Frequency of Patients With Maximum Time-Matched QT Interval (Electrocardiogram (ECG) Interval From the Beginning of the QRS Complex to the End of the T Wave) Change From Baseline Categorized by Magnitude of Change, Days 1 and 15
Description: Number of patients with maximum time-matched change from baseline in the QT interval observed at each point in time, i.e., 9 time points on Day 1 and 10 timepoints on Day 15 is reported. 3 categories of individual QTcF increases from baseline to maximum value were defined:
  <= 30 milliseconds (ms)
  > 30 to 60 milliseconds (ms)
  > 60 milliseconds (ms) Changes more than 60 ms in the QT interval represent notable changes. Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 1, 1-12 hour (h): <= 60 milliseconds (ms) | 64
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 1, 1-12 hour (h): > 60 milliseconds (ms) | 0
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: number analyzed (Participants) | 63
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: <= 60 milliseconds (ms) | 62
  Frequency of patients with maximum time-matched QTcF change from baseline on Day 15, -0:05-12 h: > 60 milliseconds (ms) | 1

28. Secondary Outcome: Number of Participants With New (Not Present at Any Time Pre-dose) Onset of QTcF ≤450 Milliseconds (ms), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula.
  Number of participants with new onset (not present at any time pre-dose) of QTcF ≤450 milliseconds (ms) on Day 1 (first drug dose nintedanib (BIBF 1120)) and Day 15 (steady state) compared to the baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) is reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Number of participants with new onset of QTcF ≤450 (ms) on Day 1 | 3
  Number of participants with new onset of QTcF ≤450 (ms) on Day 15: number analyzed (Participants) | 63
  Number of participants with new onset of QTcF ≤450 (ms) on Day 15 | 2

29. Secondary Outcome: Number of Participants With New (Not Present at Any Time Pre-dose) Onset of QTcF >450 to 470 Milliseconds (ms), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula.
  Number of participants with new onset of QTcF >450 to 470 milliseconds (ms) on Day 1 (first drug dose nintedanib (BIBF 1120)) and Day 15 (steady state) compared to the baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) is reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Number of participants with new onset of QTcF >450 to 470 ms on Day 1 | 1
  Number of participants with new onset of QTcF >450 to 470 ms on Day 15: number analyzed (Participants) | 63
  Number of participants with new onset of QTcF >450 to 470 ms on Day 15 | 1

30. Secondary Outcome: Number of Participants With New Onset of QTcF> 470 to 500 Milliseconds (ms), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula.
  Number of participants with new onset of QTcF> 470 to 500 milliseconds (ms) on Day 1 (first drug dose nintedanib (BIBF 1120)) and Day 15 (steady state) compared to the baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) is reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Number of participants with new onset of QTcF> 470 to 500 ms on Day 1 | 0
  Number of participants with new onset of QTcF> 470 to 500 ms on Day 15 | 1

31. Secondary Outcome: Number of Participants With New (Not Present at Any Time Pre-dose) Onset of QTcF> 500 Milliseconds (ms) (Notable Prolongation), Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: QTcF interval is the QT interval (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave) corrected for the effects of heart rate (HR) by the Fridericia formula.
  Number of participants with new onset of QTcF> 500 milliseconds (ms) (notable prolongation) on Day 1 (first drug dose nintedanib (BIBF 1120)) and Day 15 (steady state) compared to the baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) is reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Number of participants with new onset of QTcF> 500 (ms) on Day 1, 1-12 hour (h) | 0
  Number of participants with new onset of QTcF> 500 (ms) (notable prolongation) on Day 15, -0:05-12 h: number analyzed (Participants) | 63
  Number of participants with new onset of QTcF> 500 (ms) (notable prolongation) on Day 15, -0:05-12 h | 0

32. Secondary Outcome: Number of Participants With New (Not Present at Any Time Pre-dose) Onset of QT (Electrocardiogram (ECG) Interval From the Beginning of the QRS Complex to the End of the T Wave) > 500 ms (Notable Prolongation), Days 1 and 15 of Treatment Cycle 1
Description: Number of participants with new onset of QT (electrocardiogram (ECG) interval from the beginning of the QRS complex to the end of the T wave)> 500 milliseconds (ms) (notable prolongation) on Day 1 (first drug dose nintedanib (BIBF 1120)) and Day 15 (steady state) compared to the baseline (Day -1 prior to the first dosing of nintedanib (BIBF 1120)) is reported.
  Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  Number of participants with new onset of QT> 500 (ms) on Day 1, 1-12 hour (h) | 0
  Number of participants with new onset of QT> 500 (ms) on Day 15, -0:05-12 h: number analyzed (Participants) | 63
  Number of participants with new onset of QT> 500 (ms) on Day 15, -0:05-12 h | 0

33. Secondary Outcome: Absolute Values at Baseline (Day -1) and Day 1 and Changes From Baseline to Day 1 at Each Point in Time in PR Interval
Description: The PR interval is an electrocardiogram (ECG) interval and is the time from the onset of the P wave to the start of the QRS complex (combination of the Q wave, R wave and S wave). It reflects conduction through the atrioventricular node (AV) node. The normal PR interval is between 120 - 200 milliseconds (ms) (0.12-0.20s) in duration. Absolute values at baseline (Day-1 prior to the first dosing of nintedanib) and at Day 1 (first drug dose of nintedanib (BIBF 1120)) and changes from baseline to Day 1 at each point in time i.e., 10 time points from 0 to 12 in the PR interval are reported.
Time Frame: At 5 minutes (min) before the first dose and at 1 hour (h), at 2 h, at 3 h, at 4 h, at 5 h, at 6 h, at 7 h, at 10 h and at 12 h after the first dose of nintedanib on Day 1. Baseline (Day -1) values were taken at exactly the same time points as on Day 1.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Absolute value in PR interval on Day -1 at -5 minutes (min) | 164.7 (23.8)
  Absolute value in PR interval on Day -1 at 1 hour (h) | 165.7 (24.9)
  Absolute value in PR interval on Day -1 at 2 h | 166.8 (24.9)
  Absolute value in PR interval on Day -1 at 3 h | 166.6 (24.0)
  Absolute value in PR interval on Day -1 at 4 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day -1 at 4 h | 168.1 (26.9)
  Absolute value in PR interval on Day -1 at 5 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day -1 at 5 h | 167.2 (26.3)
  Absolute value in PR interval on Day -1 at 6 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day -1 at 6 h | 168.1 (26.4)
  Absolute value in PR interval on Day -1 at 7 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day -1 at 7 h | 168.9 (27.5)
  Absolute value in PR interval on Day -1 at 10 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day -1 at 10 h | 168.0 (26.7)
  Absolute value in PR interval on Day -1 at 12 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day -1 at 12 h | 170.0 (29.4)
  Absolute value in PR interval on Day 1 at -5 min: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 1 at -5 min | 165.7 (25.6)
  Absolute value in PR interval on Day 1 at 1 h | 167.4 (28.2)
  Absolute value in PR interval on Day 1 at 2 h | 169.4 (28.2)
  Absolute value in PR interval on Day 1 at 3 h | 170.0 (27.3)
  Absolute value in PR interval on Day 1 at 4 h | 170.0 (28.2)
  Absolute value in PR interval on Day 1 at 5 h | 169.4 (27.5)
  Absolute value in PR interval on Day 1 at 6 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 1 at 6 h | 170.8 (27.9)
  Absolute value in PR interval on Day 1 at 7 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 1 at 7 h | 169.9 (27.0)
  Absolute value n PR interval on Day 1 at 10 h: number analyzed (Participants) | 61
  Absolute value n PR interval on Day 1 at 10 h | 169.8 (26.3)
  Absolute value in PR interval on Day 1 at 12 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day 1 at 12 h | 171.3 (28.7)
  Time-matched change from Day -1 to Day 1 in PR interval at -5 min: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 1 in PR interval at -5 min | 0.7 (7.6)
  Time-matched change from Day -1 to Day 1 in PR interval at 1 h | 1.7 (11.6)
  Time-matched change from Day -1 to Day 1 in PR interval at 2 h | 2.6 (10.3)
  Time-matched change from Day -1 to Day 1 in PR interval at 3 h | 3.4 (9.1)
  Time-matched change from Day -1 to Day 1 in PR interval at 4 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 1 in PR interval at 4 h | 2.2 (9.1)
  Time-matched change from Day -1 to Day 1 in PR interval at 5 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 1 in PR interval at 5 h | 2.8 (10.7)
  Time-matched change from Day -1 to Day 1 in PR interval at 6 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 1 in PR interval at 6 h | 3.3 (9.8)
  Time-matched change from Day -1 to Day 1 in PR interval at 7 h | 1.6 (9.3)
  Time-matched change from Day -1 to Day 1 in PR interval at 10 h: number analyzed (Participants) | 60
  Time-matched change from Day -1 to Day 1 in PR interval at 10 h | 1.8 (8.6)
  Time-matched change from Day -1 to Day 1 in PR interval at 12 h | 0.7 (9.4)

34. Secondary Outcome: Absolute Values at Baseline (Day -1) and Day 15 and Changes From Baseline to Day 15 at Each Point in Time in PR Interval
Description: The PR interval is an electrocardiogram (ECG) interval and is the time from the onset of the P wave to the start of the QRS complex (combination of the Q wave, R wave and S wave). It reflects conduction through the atrioventricular node (AV) node. The normal PR interval is between 120 - 200 milliseconds (ms) (0.12-0.20s) in duration. Absolute values at baseline (Day-1 prior to the first dosing of nintedanib (BIBF 1120) and at Day 15 (steady state) and changes from baseline to Day 15 at each point in time i.e., 10 time points from 0 to 12 in the PR interval are reported.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Absolute value in PR interval on Day -1 at -5 minutes (min): number analyzed (Participants) | 63
  Absolute value in PR interval on Day -1 at -5 minutes (min) | 164.7 (24.0)
  Absolute value in PR interval on Day -1 at 1 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day -1 at 1 h | 165.7 (25.1)
  Absolute value in PR interval on Day -1 at 2 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day -1 at 2 h | 166.8 (25.1)
  Absolute value in PR interval on Day -1 at 3 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day -1 at 3 h | 166.5 (24.2)
  Absolute value in PR interval on Day -1 at 4 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day -1 at 4 h | 168.0 (27.2)
  Absolute value in PR interval on Day -1 at 5 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day -1 at 5 h | 167.2 (26.5)
  Absolute value in PR interval on Day -1 at 6 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day -1 at 6 h | 168.3 (26.6)
  Absolute value in PR interval on Day -1 at 7 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day -1 at 7 h | 168.9 (27.7)
  Absolute value in PR interval on Day -1 at 10 h: number analyzed (Participants) | 60
  Absolute value in PR interval on Day -1 at 10 h | 168.1 (26.9)
  Absolute value in PR interval on Day -1 at 12 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day -1 at 12 h | 170.1 (29.7)
  Absolute value in PR interval on Day 15 at -5 min: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at -5 min | 164.5 (24.4)
  Absolute value in PR interval on Day 15 at 1 h: number analyzed (Participants) | 62
  Absolute value in PR interval on Day 15 at 1 h | 166.1 (25.3)
  Absolute value in PR interval on Day 15 at 2 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at 2 h | 166.8 (26.2)
  Absolute value in PR interval on Day 15 at 3 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at 3 h | 167.4 (25.3)
  Absolute value in PR interval on Day 15 at 4 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at 4 h | 168.7 (27.4)
  Absolute value in PR interval on Day 15 at 5 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at 5 h | 167.7 (27.8)
  Absolute value in PR interval on Day 15at 6 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15at 6 h | 169.3 (26.7)
  Absolute value in PR interval on Day 15 at 7 h: number analyzed (Participants) | 63
  Absolute value in PR interval on Day 15 at 7 h | 169.0 (27.9)
  Absolute value in PR interval on Day 15 at 10 h: number analyzed (Participants) | 61
  Absolute value in PR interval on Day 15 at 10 h | 169.1 (27.9)
  Absolute value in PR interval on Day 15 at 12:00 h:min: number analyzed (Participants) | 60
  Absolute value in PR interval on Day 15 at 12:00 h:min | 168.8 (27.9)
  Time-matched change from Day -1 to Day 15 in PR interval at -5 min: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in PR interval at -5 min | -0.1 (10.6)
  Time-matched change from Day -1 to Day 15 in PR interval at 1 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 15 in PR interval at 1 h | 0.5 (12.5)
  Time-matched change from Day -1 to Day 15 in PR interval at 2 h: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in PR interval at 2 h | -0.0 (12.7)
  Time-matched change from Day -1 to Day 15 in PR interval at 3 h: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in PR interval at 3 h | 0.9 (14.6)
  Time matched - change from Day -1 to Day 15 in PR interval at 4 h: number analyzed (Participants) | 61
  Time matched - change from Day -1 to Day 15 in PR interval at 4 h | 0.9 (12.2)
  Time-matched change from Day -1 to Day 15 in PR interval at 5 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 15 in PR interval at 5 h | 0.9 (13.7)
  Time-matched change from Day -1 to Day 15 in PR interval at 6 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 15 in PR interval at 6 h | 1.3 (11.8)
  Time-matched change from Day -1 to Day 15 in PR interval at 7 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 15 in PR interval at 7 h | 0.6 (13.2)
  Time-matched change from Day -1 to Day 15 in PR interval at 10 h: number analyzed (Participants) | 60
  Time-matched change from Day -1 to Day 15 in PR interval at 10 h | 1.2 (11.2)
  Time-matched change from Day -1 to Day 15 in PR interval at 12 h: number analyzed (Participants) | 60
  Time-matched change from Day -1 to Day 15 in PR interval at 12 h | -1.5 (12.5)

35. Secondary Outcome: Absolute Values at Baseline (Day -1) and Day 1 and Changes From Baseline to Day 1 at Each Point in Time in QRS Interval
Description: QRS interval is an electrocardiogram (ECG) interval and is the time interval from the onset to the end of the QRS complex (combination of the Q wave, R wave and S wave). The normal QRS duration is less than 120 milliseconds (ms). Absolute values and changes from baseline (Day-1 prior to the first dosing of nintedanib) to Day 1 (first drug dose of nintedanib (BIBF 1120)) at each point in time i.e., 10 time points from 0 to 12 in the QRS interval are reported.
Time Frame: as for outcome 33
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Absolute value in QRS interval on Day -1 at -5 minutes (min) | 92.4 (11.8)
  Absolute value in QRS interval on Day -1 at 1 h | 93.7 (11.0)
  Absolute value in QRS interval on Day -1 at 2 h | 93.2 (10.5)
  Absolute value in QRS interval on Day -1 at 3 h | 93.6 (10.8)
  Absolute value in QRS interval on Day -1 at 4 h: number analyzed (Participants) | 62
  Absolute value in QRS interval on Day -1 at 4 h | 92.7 (9.8)
  Absolute value in QRS interval on Day -1 at 5 h: number analyzed (Participants) | 62
  Absolute value in QRS interval on Day -1 at 5 h | 92.6 (11.0)
  Absolute value in QRS interval on Day -1 at 6 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day -1 at 6 h | 92.5 (10.3)
  Absolute value in QRS interval on Day -1 at 7 h: number analyzed (Participants) | 62
  Absolute value in QRS interval on Day -1 at 7 h | 93.0 (10.6)
  Absolute value in QRS interval on Day -1 at 10 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day -1 at 10 h | 92.8 (11.7)
  Absolute value in QRS interval on Day -1, 12 h: number analyzed (Participants) | 62
  Absolute value in QRS interval on Day -1, 12 h | 92.5 (10.4)
  Absolute value in QRS interval on Day 1 at -5 min: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 1 at -5 min | 92.6 (10.1)
  Absolute value in QRS interval on Day 1 at 1 h | 93.2 (11.0)
  Absolute value in QRS interval on Day 1 at 2 h | 93.0 (10.4)
  Absolute value in QRS interval on Day 1 at 3 h | 93.3 (10.3)
  Absolute value in QRS interval on Day 1 at 4 h | 93.5 (11.1)
  Absolute value in QRS interval on Day 1 at 5 h | 93.4 (11.5)
  Absolute value in QRS interval on Day 1 at 6 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 1 at 6 h | 93.4 (10.7)
  Absolute value in QRS interval on Day 1 at 7 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 1 at 7 h | 93.2 (11.3)
  Absolute value in QRS interval on Day 1 at 10 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day 1 at 10 h | 92.3 (10.6)
  Absolute value in QRS interval on Day 1 at 12 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day 1 at 12 h | 92.8 (10.9)
  Time-matched change from Day -1 to Day 1 in QRS interval at -5 min: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 1 in QRS interval at -5 min | 0.7 (5.1)
  Time-matched change from Day -1 to Day 1 in QRS interval at 1 h | -0.5 (5.2)
  Time-matched change from Day -1 to Day 1 in QRS interval 2 h | -0.2 (4.4)
  Time-matched change from Day -1 to Day 1 in QRS interval at 3h | -0.3 (4.4)
  Time-matched change from Day -1 to day 1 in QRS interval at 4 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to day 1 in QRS interval at 4 h | 0.2 (4.7)
  Time-matched change from Day -1 to Day 1 in QRS interval at 5 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 1 in QRS interval at 5 h | 0.2 (5.4)
  Time-matched change from Day -1 to Day 1 in QRS interval at 6 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 1 in QRS interval at 6 h | 0.3 (5.6)
  Time-matched change from Day -1 to Day 1 in QRS interval at 7 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 1 in QRS interval at 7 h | -0.2 (4.7)
  Time-matched change from Day -1 to Day 1 in QRS interval at 10 h: number analyzed (Participants) | 60
  Time-matched change from Day -1 to Day 1 in QRS interval at 10 h | -0.5 (4.9)
  Time-matched change from Day -1 to Day 1 in QRS interval at 12 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 1 in QRS interval at 12 h | 0.3 (4.9)

36. Secondary Outcome: Absolute Values at Baseline (Day -1) and Day 15 and Changes From Baseline to Day 15 at Each Point in Time in QRS Interval
Description: QRS interval is an electrocardiogram (ECG) interval and is the time interval from the onset to the end of the QRS complex (combination of the Q wave, R wave and S wave). The normal QRS duration is less than 120 milliseconds (ms). Absolute values and changes from baseline (Day-1 prior to the first dosing of nintedanib) to Day 15 (steady state) at each point in time i.e., 10 time points from 0 to 12 in the QRS interval are reported.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
milliseconds (ms)
  Absolute value in QRS interval on Day -1 at -5 minutes (min): number analyzed (Participants) | 63
  Absolute value in QRS interval on Day -1 at -5 minutes (min) | 92.5 (11.8)
  Absolute value in QRS interval on Day -1 at 1 hour (h): number analyzed (Participants) | 63
  Absolute value in QRS interval on Day -1 at 1 hour (h) | 93.8 (11.1)
  Absolute value in QRS interval on Day -1 at 2 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day -1 at 2 h | 93.3 (10.6)
  Absolute value in QRS interval on Day -1 at 3 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day -1 at 3 h | 93.6 (10.9)
  Absolute value in QRS interval on Day -1 at 4 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day -1 at 4 h | 92.7 (9.9)
  Absolute value in QRS interval on Day -1 at 5 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day -1 at 5 h | 92.7 (11.0)
  Absolute value in QRS interval on Day -1 at 6 h: number analyzed (Participants) | 62
  Absolute value in QRS interval on Day -1 at 6 h | 92.7 (10.3)
  Absolute value in QRS interval on Day -1 at 7 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day -1 at 7 h | 93.1 (10.6)
  Absolute value in QRS interval on Day -1 at 10 h: number analyzed (Participants) | 60
  Absolute value in QRS interval on Day -1 at 10 h | 92.8 (11.8)
  Absolute value in QRS interval on Day -1 at 12 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day -1 at 12 h | 92.6 (10.4)
  Absolute value in QRS interval on Day 15 at -5 min: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at -5 min | 93.3 (11.0)
  Absolute value Day 15, 1 h: number analyzed (Participants) | 62
  Absolute value Day 15, 1 h | 93.9 (10.3)
  Absolute value in QRS interval on Day 15 at 2 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 2 h | 93.0 (11.5)
  Absolute value in QRS interval on Day 15 at 3 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 3 h | 92.9 (11.1)
  Absolute value in QRS interval on Day 15 at 4 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 4 h | 92.6 (11.2)
  Absolute value in QRS interval on Day 15 at 5 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 5 h | 93.6 (10.9)
  Absolute value in QRS interval on Day 15 at 6 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 6 h | 93.1 (11.1)
  Absolute value in QRS interval on Day 15 at 7 h: number analyzed (Participants) | 63
  Absolute value in QRS interval on Day 15 at 7 h | 93.1 (11.3)
  Absolute value in QRS interval on Day 15 at 10 h: number analyzed (Participants) | 61
  Absolute value in QRS interval on Day 15 at 10 h | 92.8 (10.7)
  Absolute value in QRS interval on Day 15 at 12 h: number analyzed (Participants) | 60
  Absolute value in QRS interval on Day 15 at 12 h | 93.7 (11.5)
  Time-matched change from Day -1 to Day 15 in QRS interval at -5 min: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in QRS interval at -5 min | 0.8 (5.4)
  Time-matched change from Day -1 to Day 15 in QRS interval at 1 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 15 in QRS interval at 1 h | 0.0 (5.1)
  Time-matched change from Day -1 to Day 15 in QRS interval at 2 h: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in QRS interval at 2 h | -0.3 (5.3)
  Time-matched change from Day -1 to Day 15 in QRS interval at 3 h: number analyzed (Participants) | 63
  Time-matched change from Day -1 to Day 15 in QRS interval at 3 h | -0.8 (5.7)
  Time-matched change from Day -1 to Day 15 in QRS interval at 4 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 15 in QRS interval at 4 h | -0.6 (5.4)
  Time-matched change from Day -1 to Day 15 in QRS interval at 5 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 15 in QRS interval at 5 h | 0.5 (7.3)
  Time-matched change from Day -1 to Day 15 in QRS interval at 6 h: number analyzed (Participants) | 62
  Time-matched change from Day -1 to Day 15 in QRS interval at 6 h | -0.1 (5.3)
  Time-matched change from Day -1 to Day 15 in QRS interval at 7 h: number analyzed (Participants) | 61
  Time-matched change from Day -1 to Day 15 in QRS interval at 7 h | -0.4 (5.3)
  Time-matched change from Day -1 to Day 15 in QRS interval at 10 h | 0.1 (5.1)
  Time-matched change from Day -1 to Day 15 in QRS interval at 12 h | 1.0 (4.7)

37. Secondary Outcome: Frequency of Patients by Clinical Electrocardiogram (ECG) Measurement Interpretation, Calculated Separately for Days 1 and 15 of Treatment Cycle 1
Description: Based on the interpretation of the electrocardiogram (ECG) patients were classified in 3 categories:
  * Normal (a normal ECG reading would be a reading that includes the following normal findings: 1) normal general features; 2) no arrhythmia; 3) no conduction delays; 4) T-wave morphology of normal; and 5) normal U-wave morphology) on Day 1 or on Day 15)
  * Not normal and not normal at baseline (an abnormal ECG reading would be a reading that includes one or more of the following abnormal findings: 1) abnormal general features; 2) arrhythmia; 3) conduction delays; 4) T-wave morphology of flat, inverted or biphasic; and 5) abnormal U-wave morphology) on Day 1 or on Day 15)
  * Not normal and new onset of finding; Time frame: Baseline (Day -1) values were taken at exactly the same time points as on Day 15.
Time Frame: as for outcome 17
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120)
Number analyzed (Participants) | 64
Participants
  ECG interpretation on Day 1: Normal | 39
  ECG interpretation on Day 1: Not normal and not normal at baseline | 24
  ECG interpretation on Day 1: Not normal and new onset of finding | 1
  ECG interpretation on Day 15: number analyzed (Participants) | 63
  ECG interpretation on Day 15: Normal | 37
  ECG interpretation on Day 15: Not normal and not normal at baseline | 25
  ECG interpretation on Day 15: Not normal and new onset of finding | 1

38. Secondary Outcome: Frequency of Adverse Events Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3.0
Description: The number of participants who experienced adverse events graded according to NCI CTCAE version 3.0, is reported below.The maximum grade of adverse event intensity for each type of treatment-related adverse event was recorded for each patient.
  Grade 1 - Mild AE Grade 2 - Moderate AE Grade 3 - Severe AE Grade 4 - Life-threatening or disabling AE Grade 5 - Death related to AE
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Participants
  Grade 1 | 11 | 5
  Grade 2 | 16 | 6
  Grade 3 | 14 | 16
  Grade 4 | 10 | 2
  Grade 5 | 7 | 1

39. Secondary Outcome: Number of Participants With Adverse Events Leading to Dose Reduction
Description: Number of participants who experienced Adverse Events which led to dose reduction of the trial medication is reported for each treatment arm.
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Participants | 16 | 8

40. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation of Trial Drug
Description: Number of participants with Adverse Events which lead to discontinuation of trial medication drug is reported for each treatment arm.
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Participants | 11 | 5

41. Secondary Outcome: Number of Participants With Adverse Events Requiring or Prolonging Hospitalisation
Description: Number of participants who experienced Adverse Events which required or prolonged hospitalisation of patients is reported for each treatment arm.
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 32
Participants | 15 | 10

42. Secondary Outcome: Duration of Hospital Stays Due to Adverse Events Requiring or Prolonging Hospitalisation
Description: Duration of hospitalisation in days for each treatment arm is reported for those patients who experienced adverse events which required or prolonged hospitalisation (of the patients).
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment and experienced Adverse Events requiring or prolonging hospitalisation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 15 | 10
days | 11.40 (8.56) | 13.10 (8.32)

43. Secondary Outcome: Frequency of Patients With Possible Clinically Significant Abnormal Lab Values
Description: Number of patients with possible clinically significant abnormal lab values for the lab parameters alkaline phosphatase, activated partial thromboplastin time (APTT), creatinine, haemoglobin, prothrombin time (PT)-international normalized ratio (INR), potassium, lymphocytes, sodium, neutrophils, platelets, aspartate amino transferase (AST), alanine aminotransferase (ALT), bilirubin and white blood cell count is reported. Only lab values with CTCAE rule for possible clinical significance are displayed.
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Population: Treated set (TS): All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment. 1 patient in the Sunitinib arm did not have on-treatment lab values.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
Number analyzed (Participants) | 64 | 31
Participants
  Alkaline phosphatase | 2 | 3
  APTT (Activated partial thrombopl. time) | 7 | 0
  Creatinine | 4 | 5
  Haemoglobin | 6 | 6
  Prothrombin time (PT)-international normalized ratio (INR) | 5 | 0
  Potassium | 14 | 4
  Lymphocytes | 8 | 11
  Sodium | 14 | 3
  Neutrophils | 3 | 9
  Platelets | 2 | 3
  Aspartate amino Transferase (AST) | 10 | 1
  Alanine aminotransferase (ALT) | 14 | 3
  Bilirubin, total | 4 | 3
  White blood cell count | 0 | 7

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to 28 days after last dose of study drug, up to 121 months.
Description: Treated set (TS): All patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Arm/Group | Nintedanib (BIBF 1120) | Sunitinib
All-Cause Mortality (participants affected / at risk) | 50/64 | 25/32
Serious Adverse Events (participants affected / at risk) | 20/64 | 11/32
Other Adverse Events (participants affected / at risk) | 55/64 | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (BIBF 1120) (N=64) | Sunitinib (N=32)
Myocardial infarction (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Obstruction (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0
Hernia repair (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (BIBF 1120) (N=64) | Sunitinib (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 40 | 15
Dry mouth (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Flatulence (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 25 | 8
Stomatitis (Gastrointestinal disorders) | 0 | 10
Vomiting (Gastrointestinal disorders) | 10 | 6
Asthenia (General disorders) | 5 | 2
Fatigue (General disorders) | 17 | 8
Hyperthermia (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 0 | 2
Pain (General disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 5 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 1
Blood creatinine increased (Investigations) | 3 | 3
Blood thyroid stimulating hormone increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 8 | 1
Lipase increased (Investigations) | 2 | 4
Weight decreased (Investigations) | 8 | 2
Weight increased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 12 | 6
Dysgeusia (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 7 | 1
Lethargy (Nervous system disorders) | 3 | 2
Haematuria (Renal and urinary disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Aortic arteriosclerosis (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 2 | 5
Aortic valve sclerosis (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Periorbital oedema (Eye disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Amylase increased (Investigations) | 1 | 2
Blood glucose increased (Investigations) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights